CLINICAL TRIAL: NCT02421263
Title: A Randomized Controlled Trial of the Effects of Psilocybin-Facilitated Experience on the Psychology and Effectiveness of Professional Leaders in Religion
Brief Title: The Effects of Psilocybin-Facilitated Experience on the Psychology and Effectiveness of Religious Professionals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-01169
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Religious or Spiritual Problem
Keywords: Psilocybin; Pharmacologic Actions; Psychotropic Drugs
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Immediate Participation Group (Experimental): Participants will begin psilocybin intervention immediately after study enrollment.
  Interventions: Drug: Psilocybin
- Delayed Participation Group (Active Comparator): Participants will begin the psilocybin intervention 6 months after study enrollment.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Participants will receive 20 mg/70 kg of psilocybin in the first session and will receive either 20 or 30 mg/70 kg in the second session.

SUMMARY:
The current protocol is a pilot study of the effects and possible utility of psilocybin-facilitated experiences for professional religious leaders. We hypothesize that religious professionals, given their interests, training, and life experience, will be able to make nuanced discriminations of their psilocybin experiences, thus contributing to the scientific understanding of mystical-type experience. As we better characterize the phenomenology of psilocybin-induced mystical experiences, we may apply this knowledge to improve potential treatment studies in the future. A primary objective is to investigate changes in psychological functioning, spirituality, health, well-being, prosocial attitudes and behavior in professional religious leaders that may occur after receiving psilocybin under supportive conditions. A secondary objective is to determine whether participants who report having had the strongest mystical-type effects during psilocybin sessions will show the largest positive changes in the Interim Questionnaire.

DETAILED DESCRIPTION:
This randomized-controlled pilot study uses a wait-list control design. A wait-list design includes a control group that is assigned to a waiting list to receive an intervention after the active treatment group does. In this study, the active group will receive the psilocybin at weeks 5 and 9 and the wait-list control group will receive psilocybin at weeks 30 and 34. The wait-list control group serves the purpose of providing an untreated comparison for the active treatment group, while at the same time allowing the wait-list participants an opportunity to obtain the intervention at a later date.

This study's procedures include screening, preparatory meetings, psilocybin sessions, and follow-up assessments. A large battery of behavioral and psychological measures will be assessed throughout. The study team will consent and enroll up to 86 subjects to obtain a total of 12 completer participants as well as 2-3 family members or friends per study participant who can assess said completers on the Observer Rating Form (COM-R). This number will account for screen-failures and dropouts as well. The 12 participants will be randomly assigned to either an immediate participation group (N=6) or a 6-month delayed participation group (N=6). Although statistical power calculations show that 12 participants will be sufficient to detect the major effects anticipated in this study, the sponsor of this study (The Council on Spiritual Practices) is concurrently funding Johns Hopkins University School of Medicine to conduct a methodologically identical study with 12 additional participants (IND #59009). This will permit the two sites to collaborate post study completion and combine the data from the two studies to provide statistical power to detect even more subtle effects of the psilocybin intervention. Twelve volunteers (6 from each group) will participate at Johns Hopkins and 12 at New York University. Randomization and data analysis will be conducted at New York University.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for religious professionals:

  * 25 to 76 years old
  * Have given written informed consent
  * College graduation or equivalent and graduate/professional training.
  * Recognized leadership position in a well-established religious organization; professional activities must include significant time interacting with those seeking religious/spiritual guidance or support.
  * During the next two years there is no foreseen likelihood for a major potentially life-altering event for her or himself or a close family member (e.g. retirement or major career change for the volunteer; life-threatening illness of a spouse or child of the volunteer)
  * Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of psilocybin session days. If the participant does not routinely consume caffeinated beverages, he/she must agree not to do so on session days.
  * Agree to refrain from using any psychoactive drugs, including alcoholic beverages and nicotine, 24 hours before and after each drug administration. The exception is caffeine. Participants will be required to be either a non-smoker or a non-daily smoker.
  * Agree not to take any PRN medications on the mornings of drug sessions
  * Agree not to take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours of each drug administration.
  * Agree that for one week before each drug session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.
  * Have no or limited lifetime use of hallucinogens. Preference will be given to enrolling volunteers with no prior use. If we decide to enroll a volunteer with prior use, preference will be given for those who report the fewest exposures or the least enduring effects from such use.

Exclusion Criteria:

* General medical exclusion criteria for religious professionals:

  * Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child-bearing potential and sexually active who are not practicing an effective means of birth control.
  * Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., symptomatic atrial fibrilation), or TIA in the past year
  * Epilepsy with history of seizures
  * Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
  * Currently taking psychoactive prescription medication on a regular (e.g., daily) basis
  * Currently taking on a regular (e.g., daily) basis any medications having a primary centrally-acting pharmacological effect on serotonin neurons or medications that are MAO inhibitors. For individuals who have intermittent or PRN use of such medications, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
  * More than 20% outside the upper or lower range of ideal body weight according to Metropolitan Life height and weight table

Psychiatric Exclusion Criteria for religious professionals:

* Current or past history of meeting DSM-5 criteria for Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I or II Disorder
* Current or past history within the last 5 years of meeting DSM-5 criteria for alcohol or substance use disorder (excluding caffeine and nicotine) or severe major depression
* Have a first or second-degree relative with Schizophrenia, Psychotic Disorder (unless substance induced or due to a medical condition), or Bipolar I or II Disorder
* Has a psychiatric condition judged to be incompatible with establishment of rapport or safe exposure to psilocybin
* History of violent or suicidal behavior
* Family history of completed suicide

Ages: 25 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Interim Questionnaire | 6-Months after enrollment
  This questionnaire asks about experiences and changes in attitudes, mood and behavior that occurred during the past 5 months. The questionnaire includes questions about salient spiritual experiences, changes in spiritual practices, changes in attitudes, moods, social interactions, and other behaviors related to participants' religious/spiritual vocation.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bossis, PhD, Study Director — New York University; Stephen Ross, MD, Principal Investigator — New York University
Locations (1):
- NYU Langone Medical Center/Tisch Hospital, New York, New York, United States